CLINICAL TRIAL: NCT04755283
Title: A Multicenter, RandomiZed, Active-ControLled Study to Evaluate the Safety and Tolerability of Two Blinded Doses of Abelacimab (MAA868) Compared With Open-Label Rivaroxaban in Patients With Atrial Fibrillation (AZALEA)
Brief Title: Safety and Tolerability of Abelacimab (MAA868) vs. Rivaroxaban in Patients With Atrial Fibrillation
Acronym: AZALEA-TIMI 71
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anthos Therapeutics, Inc. (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ANT-006; 2020-004507-13 (EudraCT Number); CMAA868A2204 (Other: Novartis)
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Atrial Fibrillation (AF); Stroke
Keywords: randomized; prospective; blinded endpoint evaluation; abelacimab; MAA868; rivaroxaban; atrial fibrillation; Factor XI; stroke; bleeding events; anti-coagulant; anticoagulation therapy
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — abelacimab; MAA868; Rivaroxaban

STUDY DESIGN:
Intervention Model Description: This is an event-driven, randomized, active-controlled, blinded endpoint, parallel-group study to evaluate the effect of two blinded doses of abelacimab relative to open-label rivaroxaban on the rate of major or clinically relevant non-major (CRNM) bleeding events in patients with atrial fibrillation (AF) who are at moderate-to-high risk of stroke.
Who Masked: Participant, Care Provider, Investigator
Masking Description: All care providers are blinded with the exception of the pharmacist and study team member assigned to administer the subcutaneous injection of abelacimab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Abelacimab 90 mg (MAA868) (Experimental): Treatment group 1: Abelacimab low dose subcutaneous (s.c.) monthly
  Extension Treatment Group: Abelacimab high dose subcutaneous (s.c.) monthly
  Interventions: Biological: Abelacimab
- Abelacimab 150 mg (MAA868) (Experimental): Treatment group 2: Abelacimab high dose subcutaneous (s.c.) monthly
  Extension Treatment Group: Abelacimab high dose subcutaneous (s.c.) monthly
  Interventions: Biological: Abelacimab
- Rivaroxaban (Active Comparator): Treatment group 3: Rivaroxaban 20 mg by mouth; orally (p.o.) once per day with the evening meal
  Patients with a Creatinine Clearance (CrCl) ≤50 ml/min by the Cockcroft-Gault equation will have a dose adaptation to rivaroxaban 15 mg p.o. daily.
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Biological: Abelacimab — Abelacimab provided as liquid in vial (150 mg/mL)
  Other Names: MAA868
  Arms: Abelacimab 150 mg (MAA868); Abelacimab 90 mg (MAA868)
Drug: Rivaroxaban — Rivaroxaban 15 mg and 20 mg provided as commercially available film-coated tablets
  Arms: Rivaroxaban

SUMMARY:
The purpose of the ANT-006 study is to evaluate the bleeding profile of abelacimab relative to rivaroxaban in patients with atrial fibrillation (AF) at moderate-to-high risk of stroke.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 55 years old
* Patients with a history of atrial fibrillation (AF) or atrial flutter with planned indefinite anticoagulation
* Patients with a CHA2DS2-VASc of ≥4 OR a CHA2DS2-VASc of ≥3 with at least 1 of the following:

  1. Planned concomitant use of antiplatelet medication use (i.e., aspirin and/or P2Y12 inhibitor) for the duration of the trial
  2. Creatinine Clearance (CrCl) ≤50 ml/min by the Cockcroft-Gault equation

Exclusion Criteria:

* History of hypersensitivity to any of the study drugs (including rivaroxaban) or its excipients, to drugs of similar chemical classes, or any contraindication listed in the label for rivaroxaban
* Patients with an intracranial or intraocular bleed within the 3 months prior to screening
* Clinically significant mitral stenosis (valve area <1.5 cm2)
* Mechanical heart valve or other indication for anticoagulation therapy other than atrial fibrillation (e.g., venous thromboembolism)
* Known presence of an atrial myxoma or left ventricular thrombus
* History of left atrial appendage closure or removal
* Active endocarditis

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1287 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2028-12-29 (Estimated)

CONTACTS AND LOCATIONS:
Locations (83):
- United States (28):
  - Anthos Investigative Site, Huntsville, Alabama
  - Anthos Investigative Site, Mobile, Alabama
  - Anthos Investigative Site, Stamford, Connecticut
  - Anthos Investigative Site, Clearwater, Florida
  - Anthos Investigative Site, Daytona Beach, Florida
  - Anthos Investigative Site, Largo, Florida
  - Anthos Investigative Site, Safety Harbor, Florida
  - Anthos Investigative Site, Saint Augustine, Florida
  - Anthos Investigative Site, Johns Creek, Georgia
  - Anthos Investigative Site, Owensboro, Kentucky
  - Anthos Investigative Site, Baltimore, Maryland
  - Anthos Investigative Site, Salisbury, Maryland
  - Anthos Investigative Site, Framingham, Massachusetts
  - Anthos Investigative Site, Haverhill, Massachusetts
  - Anthos Investigative Site, Lansing, Michigan
  - Anthos Investigative Site, Sewell, New Jersey
  - Anthos Investigative Site, Poughkeepsie, New York
  - Anthos Investigative Site, Southampton, New York
  - Anthos Investigative Site, Lenoir, North Carolina
  - Anthos Investigative Site, Fargo, North Dakota
  - Anthos Investigative Site, Oklahoma City, Oklahoma
  - Anthos Investigative Site, Camp Hill, Pennsylvania
  - Anthos Investigative Site, Kingsport, Tennessee
  - Anthos Investigative Site, Kingwood, Texas
  - Anthos Investigative Site, Odessa, Texas
  - Anthos Investigative Site, Tomball, Texas
  - Anthos Investigative Site, Falls Church, Virginia
  - Anthos Investigative Site, Manassas, Virginia
- Canada (5):
  - Anthos Investigative Site, Cambridge, Ontario
  - Anthos Investigative Site, Greater Sudbury, Ontario
  - Anthos Investigative Site, Oshawa, Ontario
  - Anthos Investigative Site, Greenfield Park, Quebec
  - Anthos Investigative Site, Montreal, Quebec
- Czechia (13):
  - Anthos Investigative Site, Brandýs nad Labem, Central Bohemia
  - Anthos Investigative Site, Poděbrady, Central Bohemia
  - Anthos Investigative Site, Příbram, Central Bohemia
  - Anthos Investigative Site, Slaný, Central Bohemia
  - Anthos Investigative Site, Mariánské Lázně, KA
  - Anthos Investigative Site, Trutnov, KR
  - Anthos Investigative Site, Liberec, LB
  - Anthos Investigative Site, Česká Lípa, LI
  - Anthos Investigative Site, Liberec, LI
  - Anthos Investigative Site, Pardubice, PA
  - Anthos Investigative Site, Prague, PR
  - Anthos Investigative Site, Kroměříž, ZL
  - Anthos Investigative Site, Holešov, Zlín
- Hungary (11):
  - Anthos Investigative Site, Orosháza, BE
  - Anthos Investigative Site, Baja, BK
  - Anthos Investigative Site, Budapest, BP
  - Anthos Investigative Site, Budapest, BU
  - Anthos Investigative Site, Székesfehérvár, FE
  - Anthos Investigative Site, Debrecen, HB
  - Anthos Investigative Site, Kaposvár, SO
  - Anthos Investigative Site (4002), Nyíregyháza, SZ
  - Anthos Investigative Site (4003), Nyíregyháza, SZ
  - Anthos Investigative Site, Balatonfüred, VE
  - Anthos Investigative Site, Balatonfüred, VM
- Poland (17):
  - Anthos Investigative Site, Gdynia, GDY
  - Anthos Investigative Site, Chrzanów, Lesser Poland Voivodeship
  - Anthos Investigative Site, Krakow, Lesser Poland Voivodeship
  - Anthos Investigative Site, Wroclaw, Lower Silesian Voivodeship
  - Anthos Investigative Site, Żarów, Lower Silesian Voivodeship
  - Anthos Investigative Site, Lublin, Lublin Voivodeship
  - Anthos Investigative Site, Zamość, Lubusz Voivodeship
  - Anthos Investigative Site, Płock, Masovian Voivodeship
  - Anthos Investigative Site, Warsaw, Masovian Voivodeship
  - Anthos Investigative Site, Przemyśl, Podkarpackie Voivodeship
  - Anthos Investigative Site, Gdynia, Pomeranian Voivodeship
  - Anthos Investigative Site, Bielsko-Biala, Silesian Voivodeship
  - Anthos Investigative Site, Dąbrowa Górnicza, Silesian Voivodeship
  - Anthos Investigative Site, Ruda Śląska, Silesian Voivodeship
  - Anthos Investigative Site, Tychy, Silesian Voivodeship
  - Anthos Investigative Site, Elblag, Warmian-Masurian Voivodeship
  - Anthos Investigative Site, Lodz, Łódź Voivodeship
- South Korea (3):
  - Anthos Investigative Site, Seogu, Busan
  - Anthos Investigative Site, Seongnam-si, Gyeonggi-do
  - Anthos Investigative Site, Seoul, Seoul
- Taiwan (6):
  - Anthos Investigative Site, Taipei, HSZ
  - Anthos Investigative Site, Hualien City, HUA
  - Anthos Investigative Site, Yilan, ILA
  - Anthos Investigative Site, Kaohsiung City, KHH
  - Anthos Investigative Site, Taipei, TPE
  - Anthos Investigative Site, Tiachung, TXG

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Result] Ruff CT, Patel SM, Giugliano RP, Morrow DA, Hug B, Kuder JF, Goodrich EL, Chen SA, Goodman SG, Joung B, Kiss RG, Spinar J, Wojakowski W, Weitz JI, Murphy SA, Wiviott SD, Parkar S, Bloomfield D, Sabatine MS; AZALEA-TIMI 71 Investigators. Abelacimab versus Rivaroxaban in Patients with Atrial Fibrillation. N Engl J Med. 2025 Jan 23;392(4):361-371. doi: 10.1056/NEJMoa2406674. PMID 39842011
- [Derived] Al Said S, Patel SM, Giugliano RP, Morrow DA, Goodrich EL, Murphy SA, Hug B, Parkar S, Chen SA, Goodman SG, Joung B, Kiss RG, Wojakowski W, Weitz JI, Bloomfield D, Sabatine MS, Ruff CT. Abelacimab vs Rivaroxaban in Older Individuals With Atrial Fibrillation: A Prespecified Analysis of the Phase 2b AZALEA-TIMI 71 Trial. JAMA Cardiol. 2026 Feb 4:e255418. doi: 10.1001/jamacardio.2025.5418. Online ahead of print. PMID 41637102
- [Derived] Al Said S, Patel SM, Giugliano RP, Morrow DA, Goodrich EL, Murphy SA, Hug B, Parkar S, Chen SA, Goodman SG, Joung B, Kiss RG, Wojakowski W, Weitz JI, Bloomfield D, Sabatine MS, Ruff CT. Abelacimab Versus Rivaroxaban in Patients With Atrial Fibrillation on Antiplatelet Therapy: A Prespecified Analysis of the AZALEA-TIMI 71 Trial. Circulation. 2025 Aug 5;152(5):290-296. doi: 10.1161/CIRCULATIONAHA.125.074037. Epub 2025 Jun 23. PMID 40546068

RESULTS

PARTICIPANT FLOW:
Groups:
- Abelacimab 90 mg (MAA868): Treatment group 1: Abelacimab low dose subcutaneous (s.c.) monthly Abelacimab: Abelacimab provided as liquid in vial (150 mg/mL)
- Abelacimab 150 mg (MAA868): Treatment group 2: Abelacimab high dose subcutaneous (s.c.) monthly Abelacimab: Abelacimab provided as liquid in vial (150 mg/mL)
- Rivaroxaban: Treatment group 3: Rivaroxaban 20 mg by mouth; orally (p.o.) once per day with the evening meal Participants with a Creatinine Clearance (CrCl) ≤50 ml/min by the Cockcroft-Gault equation will have a dose adaptation to rivaroxaban 15 mg p.o. daily. Rivaroxaban: Rivaroxaban 15 mg and 20 mg provided as commercially available film-coated tablets
Period: Overall Study
Arm/Group | Abelacimab 90 mg (MAA868) | Abelacimab 150 mg (MAA868) | Rivaroxaban
Started | 427 | 430 | 430
Entered Open-Label | 250 | 240 | 215
Completed | 382 | 391 | 389
Not Completed | 45 | 39 | 41
Not completed — Withdrawal by Subject | 14 | 3 | 6
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Death | 31 | 36 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abelacimab 90 mg (MAA868) | Abelacimab 150 mg (MAA868) | Rivaroxaban | Total
Number analyzed (Participants) | 427 | 430 | 430 | 1287
Age, Customized [Count of Participants; unit: Participants]
  ≥ 80 years | 87 | 81 | 90 | 258
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female sex | 195 | 193 | 184 | 572
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race was reported by the participant.
  Participants
    White | 404 | 410 | 404 | 1218
    Asian | 20 | 15 | 24 | 59
    Black | 3 | 5 | 2 | 10
Median Age [Median (Inter-Quartile Range); unit: years] | 75 [69 to 79] | 74 [69 to 78] | 74 [69 to 79] | 74 [69 to 78]
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 126 | 106 | 103 | 335
  Europe | 282 | 309 | 305 | 896
  Asia | 19 | 15 | 22 | 56
Median body-mass index (IQR) [Median (Inter-Quartile Range); unit: kg/m²] — The body-mass index is the weight in kilograms divided by the square of the height in meters. Data were missing for one participant in the 150-mg abelacimab group.
  kg/m² | 29.5 [26.0 to 33.6] | 30.0 [26.7 to 34.5] | 30.3 [27.0 to 34.4] | 29.9 [26.6 to 34.2]
Creatinine clearance ≤50 ml/min [Count of Participants; unit: Participants] — Population: The number analyzed reflects the available data for this characteristic rather than the total number of randomized participants, resulting in varying denominators.
  Participants
    number analyzed (Participants) | 425 | 430 | 429 | 1284
    (all) | 86 | 90 | 88 | 264
Pattern of atrial fibrillation [Count of Participants; unit: Participants] — Population: The number analyzed reflects the available data for this characteristic rather than the total number of randomized participants, resulting in varying denominators.
  Participants
    First detected or paroxysmal: number analyzed (Participants) | 426 | 424 | 428 | 1278
    First detected or paroxysmal | 224 | 220 | 225 | 669
    Persistent or long-standing persistent: number analyzed (Participants) | 426 | 424 | 428 | 1278
    Persistent or long-standing persistent | 87 | 84 | 97 | 268
    Permanent: number analyzed (Participants) | 426 | 424 | 428 | 1278
    Permanent | 115 | 120 | 106 | 341
Median CHA₂DS₂-VASc score [Median (Inter-Quartile Range); unit: score] — CHA₂DS₂-VASc scores range from 0 to 9, with higher scores indicating a greater risk of stroke. Congestive heart failure, hypertension, age of 65 to 74 years, diabetes, vascular disease, and female sex are each assigned 1 point; age of 75 years or older, previous stroke, transient ischemic attack, and previous thromboembolism are each assigned 2 points.
  score | 5.0 [4.0 to 5.0] | 5.0 [4.0 to 5.0] | 5.0 [4.0 to 6.0] | 5.0 [4.0 to 5.0]
CHA₂DS₂-VASc score [Count of Participants; unit: Participants] — CHA2DS2-VASc scores range from 0 to 9, with higher scores indicating a greater risk of stroke. Congestive heart failure, hypertension, age of 65 to 74 years, diabetes, vascular disease, and female sex are each assigned 1 point; age of 75 years or older, previous stroke, transient ischemic attack, and previous thromboembolism are each assigned 2 points.
  Participants
    ≤4 | 191 | 213 | 186 | 590
    5 | 135 | 131 | 130 | 396
    ≥6 | 101 | 86 | 114 | 301
Median HAS-BLED score [Median (Inter-Quartile Range); unit: score] — Modified HAS-BLED scores range from 0 to 8, with higher scores indicating a greater risk of bleeding. Hypertension, abnormal renal function, abnormal liver function, previous stroke, predisposition to bleeding, labile international normalized ratio (not assessed in this trial, so no points assigned for this variable), age greater than 65 years, concomitant use of aspirin or nonsteroidal antiinflammatory drugs, and excessive alcohol use are each assigned 1 point.
  score | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0] | 3.0 [2.0 to 3.0] | 3.0 [2.0 to 3.0]
HAS-BLED score ≥3 [Count of Participants; unit: Participants] — Modified HAS-BLED scores range from 0 to 8, with higher scores indicating a greater risk of bleeding. Hypertension, abnormal renal function, abnormal liver function, previous stroke, predisposition to bleeding, labile international normalized ratio (not assessed in this trial, so no points assigned for this variable), age greater than 65 years, concomitant use of aspirin or nonsteroidal antiinflammatory drugs, and excessive alcohol use are each assigned 1 point.
  Participants | 210 | 213 | 225 | 648
Hypertension [Count of Participants; unit: Participants] | 410 | 417 | 418 | 1245
Diabetes [Count of Participants; unit: Participants] | 223 | 231 | 245 | 699
Heart failure [Count of Participants; unit: Participants] | 192 | 182 | 206 | 580
Coronary artery disease [Count of Participants; unit: Participants] | 218 | 199 | 205 | 622
Previous ischemic stroke [Count of Participants; unit: Participants] — Population: The number analyzed reflects the available data for this characteristic rather than the total number of randomized participants, resulting in varying denominators.
  Participants
    number analyzed (Participants) | 427 | 430 | 429 | 1286
    (all) | 57 | 59 | 75 | 191
Previous transient ischemic attack [Count of Participants; unit: Participants] — Population: The number analyzed reflects the available data for this characteristic rather than the total number of randomized participants, resulting in varying denominators.
  Participants
    number analyzed (Participants) | 426 | 429 | 429 | 1284
    (all) | 38 | 25 | 32 | 95
History of bleeding [Count of Participants; unit: Participants] — Population: The number analyzed reflects the available data for this characteristic rather than the total number of randomized participants, resulting in varying denominators.
  Participants
    Any bleeding: number analyzed (Participants) | 424 | 425 | 427 | 1276
    Any bleeding | 29 | 34 | 36 | 99
    Gastrointestinal bleeding: number analyzed (Participants) | 427 | 428 | 428 | 1283
    Gastrointestinal bleeding | 16 | 22 | 23 | 61
Anticoagulation ≥60 days [Count of Participants; unit: Participants] — Population: The number analyzed reflects the available data for this characteristic rather than the total number of randomized participants, resulting in varying denominators.
  Participants
    Anticoagulation ≥60 days: number analyzed (Participants) | 426 | 430 | 430 | 1286
    Anticoagulation ≥60 days | 389 | 389 | 404 | 1182
    Vitamin K antagonist: number analyzed (Participants) | 426 | 430 | 430 | 1286
    Vitamin K antagonist | 125 | 130 | 130 | 385
    Direct oral anticoagulant: number analyzed (Participants) | 426 | 430 | 430 | 1286
    Direct oral anticoagulant | 283 | 271 | 291 | 845
    Parenteral agent: number analyzed (Participants) | 426 | 430 | 430 | 1286
    Parenteral agent | 3 | 9 | 6 | 18
    Previous use of >1 anticoagulant: number analyzed (Participants) | 426 | 430 | 430 | 1286
    Previous use of >1 anticoagulant | 22 | 21 | 23 | 66
Planned concomitant antiplatelet medication [Count of Participants; unit: Participants] — Population: The number of participants with planned concomitant antiplatelet medication are presented.
  Participants
    Aspirin: number analyzed (Participants) | 107 | 105 | 106 | 318
    Aspirin | 72 | 70 | 58 | 200
    P2Y12 inhibitor: number analyzed (Participants) | 107 | 105 | 106 | 318
    P2Y12 inhibitor | 26 | 29 | 42 | 97
    Dual antiplatelet therapy: number analyzed (Participants) | 107 | 105 | 106 | 318
    Dual antiplatelet therapy | 9 | 6 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of the First Occurrence of Composite of International Society on Thrombosis and Haemostasis (ISTH)-Defined Major Bleeding or Clinically Relevant Non-Major (CRNM) Bleeding Events
Description: The number of participants experiencing the first occurrence of the composite of ISTH-defined major bleeding or CRNM bleeding events divided by the number of 100 person-years through the first event or end of treatment across all participants, is presented. For participants not experiencing events, person-years is calculated through the end of treatment during the randomized phase.
Time Frame: Assessed at every visit from randomization through the end of the randomized phase of the study, up to 33 months.
Population: The analysis population is the number of randomized participants who received at least one dose of study treatment. The difference between the overall number of participants analyzed and the overall number of participants assigned to the arm represents those who never received a dose of study treatment.
Measure: Number; unit: participants with event/100 person-years
Arm/Group | Abelacimab 90 mg (MAA868) | Abelacimab 150 mg (MAA868) | Rivaroxaban
Number analyzed (Participants) | 425 | 427 | 428
participants with event/100 person-years | 2.64 | 3.22 | 8.39
Statistical Analysis 1: Comparison: Abelacimab 90 mg (MAA868) vs Rivaroxaban; Test type: Superiority; p < 0.001, Stratified Log Rank Test; Stratified for stratification factors; Hazard Ratio (HR) = 0.314, 95% CI 2-sided [0.192 to 0.513] — Cox Proportional Hazards Model Adjusted for Stratification Factors
Statistical Analysis 2: Comparison: Abelacimab 150 mg (MAA868) vs Rivaroxaban; Test type: Superiority; p < 0.001, Stratified Log Rank Test; Stratified for stratification factors; Hazard Ratio (HR) = 0.382, 95% CI 2-sided [0.243 to 0.602] — Cox Proportional Hazards Model Adjusted for Stratification Factors

2. Secondary Outcome: Incidence Rate of the First Occurrence of ISTH-defined Major Bleeding Events
Description: The number of participants experiencing the first occurrence of ISTH-defined major bleeding events divided by the number of 100 person-years through the first event or end of treatment across all participants, is presented. For participants not experiencing events, person-years is calculated through the end of treatment during the randomized phase.
Time Frame: Assessed at every visit from randomization through the end of the randomized phase of the study, up to 33 months.
Population: as for outcome 1
Measure: Number; unit: participants with event/100 person-years
Arm/Group | Abelacimab 90 mg (MAA868) | Abelacimab 150 mg (MAA868) | Rivaroxaban
Number analyzed (Participants) | 425 | 427 | 428
participants with event/100 person-years | 0.99 | 1.22 | 3.73
Statistical Analysis 1: Comparison: Abelacimab 90 mg (MAA868) vs Rivaroxaban; Test type: Superiority; p < 0.001, Stratified Log Rank Test; Stratified for stratification factors; Hazard Ratio (HR) = 0.263, 95% CI 2-sided [0.121 to 0.572] — Cox Proportional Hazards Model Adjusted for Stratification Factors
Statistical Analysis 2: Comparison: Abelacimab 150 mg (MAA868) vs Rivaroxaban; Test type: Superiority; p = 0.001, Stratified Log Rank Test; Stratified for stratification factors; Hazard Ratio (HR) = 0.325, 95% CI 2-sided [0.159 to 0.663] — Cox Proportional Hazards Model Adjusted for Stratification Factors

3. Secondary Outcome: Incidence Rate of the First Occurrence of ISTH-defined Major or CRNM or Minor Bleeding Events
Description: The number of participants experiencing the first occurrence of the composite of ISTH-defined major or CRNM or minor bleeding events divided by the number of 100 person-years through the first event or end of treatment across all participants, is presented. For participants not experiencing events, person-years is calculated through the end of treatment during the randomized phase.
Time Frame: Assessed at every visit from randomization through the end of the randomized phase of the study, up to 33 months.
Population: as for outcome 1
Measure: Number; unit: participants with event/100 person-years
Arm/Group | Abelacimab 90 mg (MAA868) | Abelacimab 150 mg (MAA868) | Rivaroxaban
Number analyzed (Participants) | 425 | 427 | 428
participants with event/100 person-years | 7.05 | 10.43 | 15.30
Statistical Analysis 1: Comparison: Abelacimab 90 mg (MAA868) vs Rivaroxaban; Test type: Superiority; p < 0.001, Stratified Log Rank Test; Stratified for stratification factors; Hazard Ratio (HR) = 0.460, 95% CI 2-sided [0.332 to 0.638] — Cox Proportional Hazards Model Adjusted for Stratification Factors
Statistical Analysis 2: Comparison: Abelacimab 150 mg (MAA868) vs Rivaroxaban; Test type: Superiority; p = 0.010, Stratified Log Rank Test; Stratified for stratification factors; Hazard Ratio (HR) = 0.683, 95% CI 2-sided [0.512 to 0.912] — Cox Proportional Hazards Model Adjusted for Stratification Factors

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) that started during or after the start of the treatment or started prior to the start of the treatment and increased in severity after the start of the treatment through each participant's derived End of Study date for the randomized period (up to 33 months).
Description: The appearance or worsening of any undesirable sign, symptom, or medical condition occurring after starting study drug even if event is not considered to be related to study drug is considered an AE. Reports of intentional misuse and abuse of study treatment are considered AEs, even without a clinical event. AEs may be detected by non-directive questioning, voluntary reports, or findings from exams, lab tests, or other assessments. AEs are presented for the Analysis Population.
Arm/Group | Abelacimab 90 mg (MAA868) | Abelacimab 150 mg (MAA868) | Rivaroxaban
All-Cause Mortality (participants affected / at risk) | 31/427 | 36/430 | 34/430
Serious Adverse Events (participants affected / at risk) | 158/425 | 157/427 | 167/428
Other Adverse Events (participants affected / at risk) | 215/425 | 257/427 | 227/428
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abelacimab 90 mg (MAA868) (N=425) | Abelacimab 150 mg (MAA868) (N=427) | Rivaroxaban (N=428)
Pneumonia (Infections and infestations) | 10 (11) | 10 (11) | 13 (15)
COVID-19 pneumonia (Infections and infestations) | 9 (9) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 5 (5) | 3 (3) | 5 (5)
Urinary tract infection (Infections and infestations) | 4 (4) | 7 (7) | 1 (2)
COVID-19 (Infections and infestations) | 5 (5) | 2 (2) | 3 (3)
Cellulitis (Infections and infestations) | 4 (7) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Septic shock (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Citrobacter sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Keratouveitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulvitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hormone receptor positive breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Intestinal metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Meningionma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (18)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Non-small cell lung cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 11 (13)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Bone marrow disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Pernicious anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic complication (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 6 (6) | 4 (5) | 3 (4)
Transient ischaemic attack (Nervous system disorders) | 6 (6) | 3 (3) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 4 (4) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Embolic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Axonal and demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Basal ganglia stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dementia with Lewy bodies (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Essential tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Focal dyscognitive seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Intracranial mass (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Middle cerebral artery stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vitreoretinal traction syndrome (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 26 (38) | 20 (23) | 18 (32)
Atrial fibrillation (Cardiac disorders) | 18 (27) | 14 (18) | 10 (12)
Acute myocardial infarction (Cardiac disorders) | 6 (6) | 3 (3) | 7 (9)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 6 (6) | 6 (11)
Coronary artery disease (Cardiac disorders) | 5 (5) | 2 (2) | 4 (4)
Angina unstable (Cardiac disorders) | 3 (3) | 3 (3) | 4 (4)
Cardiac failure chronic (Cardiac disorders) | 4 (4) | 3 (3) | 3 (3)
Myocardial infarction (Cardiac disorders) | 3 (4) | 1 (1) | 4 (4)
Angina pectoris (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (2) | 3 (3)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 2 (2) | 3 (5)
Sinus node dysfunction (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 3 (4)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic left ventricular failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chronotropic incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 3 (3) | 1 (1) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 3 (3) | 1 (2) | 2 (5)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 3 (3) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral vascular haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 2 (3) | 6 (9)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 3 (3) | 5 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1) | 2 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epiglottis dysfunction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3) | 12 (14)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (4) | 2 (3)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (4)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bowel movement irregularity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enterocele (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Biliary dilatation (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholestatis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (3)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Angiodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Scar discomfort (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (5) | 1 (2) | 6 (6)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 4 (4)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 9 (9) | 4 (4) | 6 (6)
Sudden cardiac death (General disorders) | 2 (2) | 4 (4) | 2 (2)
Sudden death (General disorders) | 0 (0) | 1 (1) | 3 (3)
Asthenia (General disorders) | 1 (1) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Granuloma (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Necrosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Stent-graft endoleak (General disorders) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (3)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Near drowning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 1 (1) | 0 (0)
Lead dislodgement (Product Issues) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abelacimab 90 mg (MAA868) (N=425) | Abelacimab 150 mg (MAA868) (N=427) | Rivaroxaban (N=428)
COVID-19 (Infections and infestations) | 41 (42) | 48 (49) | 45 (46)
Atrial fibrillation (Cardiac disorders) | 28 (39) | 27 (34) | 24 (31)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (26) | 26 (31) | 27 (29)
Hypertension (Vascular disorders) | 24 (25) | 26 (27) | 20 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (21) | 26 (29) | 22 (24)
Urinary tract infection (Infections and infestations) | 27 (38) | 24 (27) | 12 (12)
Anaemia (Blood and lymphatic system disorders) | 18 (23) | 17 (18) | 24 (29)
Contusion (Injury, poisoning and procedural complications) | 10 (15) | 27 (36) | 15 (19)
Headache (Nervous system disorders) | 13 (15) | 27 (33) | 11 (14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 9 (12) | 27 (41)

LIMITATIONS AND CAVEATS:
The independent data monitoring committee recommended early termination of the trial on September 14, 2023.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication by Institution or Investigator until after publication of the results by Sponsor. If there is no multicenter publication within 18 months after the end of the Study, Institution and Investigator may publish if Sponsor is given the opportunity to review at least 45 days prior to submission for publication. Sponsor may remove any Information other than Study Data from a proposed publication. Sponsor may defer publication or other disclosure for a period of 60 additional days.

DOCUMENTS (2):
  • Study Protocol (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT04755283/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/83/NCT04755283/SAP_001.pdf